CLINICAL TRIAL: NCT01237067
Title: A Pharmacokinetic/Pharmacodynamic Study With a Phase I Run-In With a PARP Inhibitor (Olaparib) in Combination With Carboplatin for Refractory or Recurrent Women's Cancers
Brief Title: Olaparib in Combination With Carboplatin for Refractory or Recurrent Women s Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110022; 11-C-0022
Record Dates: First submitted 2010-11-06; First posted 2010-11-09 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2019-12-12

CONDITIONS: Ovarian Cancer; Breast Cancer; Primary Peritoneal Cancer; Fallopian Tube Cancer; Endometrial Cancer
Keywords: PARP inhibitor, womens's cancers, relapsed, recurrent; Ovarian, breast, endometrial, cervical; Carboplatin; BRCA 1 and BRCA 2
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms; Fallopian Tube Neoplasms; Endometrial Neoplasms; Recurrence | interventions — Carboplatin; olaparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Dose esc: A phase I 3 + 3 safety run-in will optimize tablet olaparib dose (d1-7) in combination with carboplatin on day 1. The carboplatin dose through the randomized portion of the trial will be AUC4. Subsequent accrual will randomize patients to one of 2 schedules on cycle 1 with the other schedule on cycle 2. A: olaparib d1-7 > carbo d8; B: carbo d1 > olaparib d2-8. Cycle 3-8 will be schedule B. After 8 cycles of carboplatin, olaparib will be administered alone on a daily basis
  Interventions: Drug: Carboplatin; Drug: Olaparib
- Group 2A (Experimental): Randomized: A phase I 3 + 3 safety run-in will optimize tablet olaparib dose (d1-7) in combination with carboplatin on day 1. The carboplatin dose through the randomized portion of the trial will be AUC4. Subsequent accrual will randomize patients to one of 2 schedules on cycle 1 with the other schedule on cycle 2. A: olaparib d1-7 > carbo d8; B: carbo d1 > olaparib d2-8. Cycle 3-8 will be schedule B. After 8 cycles of carboplatin, olaparib will be administered alone on a daily basis.
  Interventions: Drug: Carboplatin; Drug: Olaparib
- Group 2B (Experimental): Randomized: A phase I 3 + 3 safety run-in will optimize tablet olaparib dose (d1-7) in combination with carboplatin on day 1. The carboplatin dose through the randomized portion of the trial will be AUC4. Subsequent accrual will randomize patients to one of 2 schedules on cycle 1 with the other schedule on cycle 2. A: olaparib d1-7 > carbo d8; B: carbo d1 > olaparib d2-8. Cycle 3-8 will be schedule B. After 8 cycles of carboplatin, olaparib will be administered alone on a daily basis.
  Interventions: Drug: Carboplatin; Drug: Olaparib

INTERVENTIONS:
Drug: Carboplatin — A phase I 3 + 3 safety run-in will optimize tablet olaparib dose (d1-7) in combination with carboplatin on day 1. The carboplatin dose through the randomized portion of the trial will be AUC4. Subsequent accrual will randomize patients to one of 2 schedules on cycle 1 with the other schedule on cycle 2. A: olaparib d1-7 > carbo d8; B: carbo d1 > olaparib d2-8. Cycle 3-8 will be schedule B. After 8 cycles of carboplatin, olaparib will be administered alone on a daily basis.
Drug: Olaparib — A phase I 3 + 3 safety run-in will optimize tablet olaparib dose (d1-7) in combination with carboplatin on day 1. The carboplatin dose through the randomized portion of the trial will be AUC4. Subsequent accrual will randomize patients to one of 2 schedules on cycle 1 with the other schedule on cycle 2. A: olaparib d1-7 > carbo d8; B: carbo d1 > olaparib d2-8. Cycle 3-8 will be schedule B. After 8 cycles of carboplatin, olaparib will be administered alone on a daily basis.

SUMMARY:
Background:

- Olaparib is an experimental anti-cancer drug that is part of a class of drugs called PARP inhibitors. PARP is a protein that is involved in repairing DNA damage, but it may also encourage precancerous cells to develop into cancer cells. Olaparib has been given safely in combination with carboplatin, a drug used to treat breast, ovarian, uterine, and cervical cancer, but more research is needed to determine whether the drugs are more effective when given together or which drug should be given first.

Objectives:

- To determine the safety and effectiveness of combined carboplatin and olaparib as a treatment for gynecologic (female organ) or breast cancer.

Eligibility:

* Women at least 18 years of age who have breast, ovarian, uterine, or cervical cancer that has not responded to standard treatments.
* Men at least 18 years of age who have metastatic breast cancer and have a BRCA-1/2 mutation.

Design:

* Participants will be screened with a physical examination and medical history, as well as blood and tumor samples and imaging studies as required by the researchers. Study participants will then be divided into two groups.
* Group 1: Participants will receive olaparib tablets twice a day for 7 days (14 doses) and will receive carboplatin by vein on day 1 or 2, for a 21-day treatment cycle. Group 1 study is designed to determine the safety of new tablet formulation of olaparib.
* Group 2: Participants will be divided into two smaller groups, with reversed treatment schedules. Group 2 study is designed to evaluate which drug should be given first through endpoint studies in blood samples.
* Group 2A: Participants will receive olaparib tablets twice a day for 7 days (14 doses) and then carboplatin on day 8 of the first cycle. Cycle 2 will start with carboplatin on day 1 and olaparib starting on day 2 for 7 days (14 doses).
* Group 2B: Participants will receive carboplatin on the first day of the first cycle, and then olaparib on day 2, twice a day for 7 days (14 doses) of the first cycle. Cycle 2 will start with 7 days of olaparib (14 doses) and carboplatin will be given on day 8.
* From cycle 3 until completion of therapy, all Group 2 participants will follow the schedule used for Group 1 (carboplatin on day 1 or 2 of the week of olaparib therapy, also in 21-day cycles).
* Additional blood and tissue samples and imaging studies will be conducted throughout the treatment period.
* All participants may receive no more than 8 cycles of olaparib and carboplatin therapy, but may continue to take olaparib if their cancer responds to the treatment.

DETAILED DESCRIPTION:
Background:

* Olaparib (AZD2281) is an oral PARP-1/2 inhibitor (PARPi) that affects tumors by impairing repair of single stranded DNA and causing double strand breaks. Carboplatin covalently crosslinks DNA causing stalled replication forks repaired through nucleotide excision repair and homologous recombination (HR).
* There is no published data on sequence-specificity of PARPi with platinums. Our preclinical data indicate sequence may be important in growth inhibition and DNA damage and repair.
* We have demonstrated activity and safety with concomitant administration of olaparib and carboplatin.
* We hypothesize that elucidation of sequence specificity may improve upon that clinical benefit by optimizing drug administration and potentially safety.

Objectives:

* To determine safe dose of olaparib tablet with carboplatin.
* To estimate the pharmacokinetic (PK) and pharmacodynamic (PD) effects of two schedules of olaparib and carboplatin using peripheral blood mononuclear cells (PBMCs).
* To determine the schedule-associated safety of olaparib and carboplatin in women s cancers.

Eligibility:

* Adult women with recurrent/refractory epithelial ovarian cancer, fallopian, primary peritoneal, uterine papillary serous cancer, or malignant mixed mullerian tumors, or recurrent/refractory breast cancer that is metastatic or unresectable and for which standard therapies do not exist or are no longer effective. BRCA1/2 mutation carriers will be eligible with any metastatic disease.
* Patients must be off prior chemotherapy, radiation therapy, hormonal therapy, or biological therapy for at least 4 weeks.
* ECOG performance status 0-2 and adequate organ and marrow function.

Design:

* A phase I 3 plus 3 safety run-in will optimize tablet olaparib dose (d1-7) in combination with carboplatin on day 1. The carboplatin dose through the trial will be AUC4.
* Subsequent accrual will randomize patients to one of 2 schedules on cycle 1 with the other schedule on cycle 2. A: olaparib d1-7 > carbo d8; B: carbo d1 > olaparib d2-8.
* Cycle 3-8 will be schedule B. After 8 cycles of carboplatin, olaparib will be administered alone on a daily basis.
* Research samples will be obtained for PD endpoints prior to and approximately 24 hours after carboplatin infusion and prior to the 1st and 3rd of olaparib.
* Blood samples for olaparib PK will be obtained in all patients after the first dose of olaparib in cycles 1 and 2.
* Patients will be evaluated for toxicity in clinic every 3 weeks and every two cycles for response using RECIST criteria. Imaging studies will be obtained every 3 cycles for patients who stay on the study longer than four years.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have confirmed at the NCI, histologically or cytologically recurrent/refractory gynecologic cancers such as but not restricted to epithelial ovarian, fallopian, primary peritoneal, uterine papillary serous cancer, cervix cancer, malignant mixed mullerian tumors, or any type of breast cancer that is metastatic or unresectable and for whom curative therapies do not exist.
* All patients must have measurable and/or evaluable disease; biomarker-only disease is not considered measurable or evaluable; eligibility of bone only disease is a PI decision on an individual patient basis.
* Breast cancer patients with locally advanced, unresectable disease must have been previously treated with standard therapy.
* Breast cancer patients with deleterious mutation in DNA repair enzymes with locally advanced or metastatic disease do not have to have had prior therapy for their progressive disease. Men with BRCA1/2 mutation and metastatic breast cancer will be eligible for study. Ovarian or endometrial cancer patients with deleterious mutation in DNA repair enzymes may be treated in first recurrence independent of platinum-sensitivity history.
* There is no limit on number of prior therapies. Patients must be at least 6 months from their last platinum exposure and platinum-resistant patients may participate.
* Age greater than or equal to 18 years
* ECOG performance status less than or equal to 2
* Patients must have normal organ and marrow function as defined below:

Absolute neutrophil count greater than or equal to 1,500/mm3

Platelets greater than or equal to 100,000/mm3

Serum Creatinine less or than or equal to 1.5 mg/dL or if low, Cr Cl greater than 60 mL/min

Total bilirubin less than or equal to 1.5 times the limit of normal (ULN) in the absence of Gilbert s syndrome

AST(SGOT0/ALT(SGPT) less than or equal to 3 times the ULN (CTCAE4.0 grade 2)

* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for at least three months following the last dose of experimental therapy.
* Women of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to the start of the study.
* Ability to understand and the willingness to sign a written informed consent document
* Inclusion of Women and Minorities: Women and members of all races and ethnic groups are eligible for this trial.

EXCLUSION CRITERIA:

* Patients who have had treatment for their disease, such as chemotherapy, biological therapy, radiotherapy, surgery, or complementary and alternative therapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study.
* Patients who were treated with other PARP inhibitors greater than 28 days prior to study are eligible.
* Must be at least 2 weeks from the last phase 0 intervention (longer at the discretion of the PI) and at least 1 day from non-cancer-related complementary and alternative medicine prior to entering the study.
* Previous treatment with olaparib (AZD2281).
* Invasive cancer, other than co-existent breast/gynecologic cancers, within the past 2 years. Noninvasive nonmelanoma skin cancers are not exclusions.
* Patients with known brain metastases diagnosed within 1 year will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Patients with brain metastases diagnosed greater than 1 year prior to study entry may be considered if they received sterilizing therapy to the CNS (resection or radiation) and have been CNS recurrence-free for a full 1-year period
* History of grade 4 allergic reactions to platinums:

Patients with allergic reaction to platinums (up to and including grade 3 without a reaction protocol, and up to and including grade 2 in the face of aggressive pre-treatment) may be eligible pending review of experience, and PI approval.

Patients who have not been rechallenged after a severe reaction may be eligible on a case-by-case basis.

* Clinically significant GI bleeding or hemoptysis within 28 days prior to the start of the study
* Inability to swallow pills
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (no antibiotics prior to entering the study within 7 days), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and breast-feeding women: If a woman becomes pregnant or suspects she is pregnant while participating in this study, she should inform her treating physician immediately.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with AZD2281. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy such as carboplatin. HIV- positive patients who are not on combination antiretroviral therapy but with CD4 counts >500, eligibility is a PI decision on an individual patient basis.
* Major surgery within the past 28 days

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2011-02-07; Primary Completion 2014-11-16 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Determine the pharmacodynamic effects of the sequence of administration of olaparib and carboplatin and the schedule-associated safety of the combination. | Cycle 1 at 24 and 48 hours
  Pharmacodynamic study results and toxicity during Cycle 1 at 24 and 48 hours
Safety of combination of olaparib and carboplatin | End of Cycle 2
  Toxicity at the end of Cycle 2

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Min Lee, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Alderson T. New targets for cancer chemotherapy--poly(ADP-ribosylation) processing and polyisoprene metabolism. Biol Rev Camb Philos Soc. 1990 Nov;65(4):623-41. doi: 10.1111/j.1469-185x.1990.tb01240.x. No abstract available. PMID 2124932
- [Background] Berger NA, Adams JW, Sikorski GW, Petzold SJ, Shearer WT. Synthesis of DNA and poly(adenosine diphosphate ribose) in normal and chronic lymphocytic leukemia lymphocytes. J Clin Invest. 1978 Jul;62(1):111-8. doi: 10.1172/JCI109094. PMID 659624
- [Background] Cottet F, Blanche H, Verasdonck P, Le Gall I, Schachter F, Burkle A, Muiras ML. New polymorphisms in the human poly(ADP-ribose) polymerase-1 coding sequence: lack of association with longevity or with increased cellular poly(ADP-ribosyl)ation capacity. J Mol Med (Berl). 2000;78(8):431-40. doi: 10.1007/s001090000132. PMID 11097112